CLINICAL TRIAL: NCT06064721
Title: Effect of Buerger Allen Exercise on Peripheral Circulation Among Patients With Type 2 Diabetes Mellitus Visited in Outpatients Department: A Randomized Controlled Trial
Brief Title: Effect of Buerger Allen Exercise on Peripheral Circulation Among Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Sana Zreef, principal investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PC RCT 001
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Buerger-Allen exercise and Routine care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buerger-Allen Exercise Group (Experimental): The researcher will conduct training sessions on the BAE for the study group (how to perform these exercises, duration, and frequency of exercise).
  Firstly researcher practically demonstrate the BAE technique lasting 15-20 minutes, and secondly will encourage each participant to re-demonstrate the following technique.
  The researcher will ensure that the study group practices the exercise until they demonstrate competence in its execution. Additionally, the study group will be provided with a photographic brochure illustrating the exercise.
  The buerger Allen exercise will consist of three steps step 1. Elevation step 2. Dependency step 3. Horizontal The intervention group will continue for 51 days, with a 6-8 hour gap between the two sessions, in addition to receiving routine care.
  To ensure exercise continuity, participants will receive reminders via phone calls/messages
  Interventions: Other: Buerger-Allen Exercise
- Routine Care Group (No Intervention): the control group participants will receive routine care.

INTERVENTIONS:
Other: Buerger-Allen Exercise — Buerger-Allen exercise will be taught by researcher and perform by patient at home twice a day
  Arms: Buerger-Allen Exercise Group

SUMMARY:
This randomized control trial aims to compare peripheral circulation in type 2 diabetes mellitus. This study aims to determine the effect of the Buerger-Allen exercise (BAE) on peripheral circulation among patients with type 2 diabetes mellitus visited in outpatients department Participants will perform the Buerger -Allen exercise with routine care control group: Researchers will compare with routine care

DETAILED DESCRIPTION:
Peripheral arterial disease is a common complication among patients with Type 2 diabetes mellitus (T2DM), resulting from long-term elevated blood glucose levels that damage blood vessels and impair circulation. This impaired circulation can lead to a range of complications, including poor wound healing, ulcers, and amputations. Peripheral circulation issues, particularly in the lower extremities, are of significant concern as they contribute to decreased mobility, pain, and reduced quality of life in individuals with T2DM. Buerger-Allen exercises are designed to stimulate venous return and enhance limb circulation by alternating between positions of elevation and dependency. This exercise involves different movements to increase blood flow, and improve limb function, ultimately improving quality of life. However, further research is needed to determine the precise impact of this exercise in enhancing lower extremity circulation for individuals with type 2 diabetes mellitus. This study aims to assess the effect of the Buerger-Allen exercise on peripheral circulation among patients with type 2 diabetes mellitus who visited an outpatient department. It is hypothesized that patients who will receive the Buerger-Allen exercise will have a difference in peripheral circulation than patients who will not. A randomized controlled trial will be conducted with 74 participants based on convenience sampling, randomly allocated into two groups (37 in each) through the lottery method. Recruitment for study participants will be conducted in the diabetic clinic of the outpatient department in the district headquarters hospital, Sheikhupura. Peripheral circulation will be assessed using the perfusion index, and Vascular Quality of Life Questionnaire-6 at baseline, on the 6th day, and after 15 days of the intervention. The data will be analyzed using SPSS version 27. Descriptive statistics (percentage, frequency, mean, and standard deviation) will be used to describe the characteristics of the study population. Inferential statistics such as independent t-tests and repeated measures ANOVA will be used to compare the mean score of perfusion index between both groups at different points in time, depending on the normality of data. The significance level will be set at p < 0.05. It is expected that the intervention group receiving the Buerger-Allen Exercise would demonstrate significant improvements in peripheral circulation, improving quality of life. The findings from the current study may also be substantial for physicians to recommend Buerger-Allen Exercise as adjunctive therapy in individuals with type 2 diabetes mellitus. This evidence-based intervention may also offer accessibility and reduce the need for costly hospitalizations and treatments for peripheral complications of diabetic foot, benefiting both patients and healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Type 2 diabetes mellitus
* Participants who have an age group of 35-65 years
* Participants who are using insulin for the last 5 years

Exclusion Criteria:

* Participants with a history of deep vein thrombosis
* Patients who have undergone recent surgeries on the lower extremities
* Participants with severe comorbidities, such as uncontrolled hypertension or heart failure
* Participants with cognitive impairments that hinder their ability to understand and perform the exercises safely

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2025-08-07 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
peripheral circulation | total 21 days (baseline line, 6th day, and after15th day
  peripheral circulation measure by perfusion index

CONTACTS AND LOCATIONS:
Locations (1):
- DHQ hospital, sheikhupura, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No